CLINICAL TRIAL: NCT06839222
Title: Randomized Controlled Single-Blind Multi-Centre Evaluation of the Safety and Performance of an Injection of Hydrogel OA 2% in Subjects With Knee Osteoarthritis
Brief Title: Knee OsteoArthritis Long-term Assessment
Acronym: KOALA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegro NV/SA (Industry)
Collaborators: QbD Clinical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DHF-001-DVaP-001-03
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: Hydrogel OA 2%; Knee Osteoarthritis; Knee Injury and Osteoarthritis Outcome Score (KOOS); Safety; Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Intervention Model Description: A randomized controlled, single-blind, multi-center, prospective first-inhuman clinical investigation.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrogel OA 2% (Experimental): treatment arm
  Interventions: Device: Hydrogel OA 2%
- Hyaluronic Acid (Durolane) (Active Comparator): control arm
  Interventions: Device: Hyaluronic Acid (Durolane)

INTERVENTIONS:
Device: Hydrogel OA 2% — Hydrogel OA 2% is a sterile, nonpyrogenic viscoelastic hydrogel suspension, designed using highly purified biopolymers in a phosphate-buffered saline solution. The main component is a cross-linked protein (ultra-pure bovine gelatin). The other main component is a polysaccharide cellulose nanocrystal (CNC) that acts as the crosslinker. Hydrogel OA 2% is supplied in pre-filled 2.25ml Luer lock syringe. Each package contains one syringe containing 2.0 mL Hydrogel OA 2%. Hydrogel OA 2% is designed to provide symptomatic relief by restoring joint lubrication and cushioning, potentially leading to reduced pain and improved joint function. The device is suitable for use in early and moderate OA (Kellgren and Lawrence, K&L, II-III).
  Arms: Hydrogel OA 2%
Device: Hyaluronic Acid (Durolane) — DUROLANE contains 20 mg/mL of stabilized non-animal hyaluronic acid in buffered physiological sodium chloride solution pH 7. DUROLANE is a sterile, transparent viscoelastic gel supplied in a 3 mL glass syringe.
  Arms: Hyaluronic Acid (Durolane)

SUMMARY:
The goal of this clinical study is to learn if Hydrogel OA 2% injection is safe and whether it works to improve symptoms of diagnosed knee osteoarthritis in adults when compared to Hyaluronic Acid (Durolane), a treatment that is currently often used for treatment of knee osteoarthritis. The main question it aims to answer is:

- How many study participants will experience side effects related to Hydrogel OA 2% during the study when compared to Hyaluronic Acid (Durolane)?

All study participants will receive either one Hydrogel OA 2% or Hyaluronic Acid (Durolane) injection in their knee during the clinical study. Study participants will not know which treatment they have received. Study participants will also receive a call from the researchers and visit the clinic three times to report whether they have experienced any side effects, and complete a questionnaire that will ask questions on whether their symptoms have improved since they received an injection.

ELIGIBILITY:
Inclusion Criteria:

* Adults accepting to participate in the study and having signed the written informed consent form before any protocol-specific procedures and able to understand and follow the instructions as described in the protocol.
* Unilateral symptomatic tibiofemoral KOA confirmed by a "standing knee" X-ray. In case of bilateral KOA on X-ray only one knee (indexed knee) presents symptomatic OA pain.
* Age 35 ≤ 75 years.
* BMI 20 ≤ 35.
* Knee Injury and Osteoarthritis Outcome Score (KOOS) Pain score 25-85.
* Radiological Kellgren and Lawrence (K&L) grade II and III from a standing knee radiograph with minimum joint space of 1 mm in the study knee.
* Fully ambulatory for functional assessments.
* Willingness to refrain from taking any pain medication for 48 hours prior to each study visit.
* Female subjects must be on effective contraception (pill, patch, ring, diaphragm, implant or intrauterine device), if not surgically sterile (tubal ligation or hysterectomy) or postmenopausal for at least one year. Females must show a negative pregnancy test at the treatment visit.

Exclusion Criteria:

* Bilateral tibiofemoral KOA where the non-symptomatic knee presents worse radiological grade of KOA.
* Radiological K&L grade 0, I, or IV from a standing knee radiograph assessed during the screening visit, using the most recent x-ray taken either immediately or within the past 3 months. Significant clinically assessed varus or valgus deformation of the selected knee side of more than 10 degrees.
* Extension deficit of the index knee of higher than 5 degrees.
* Bilateral symptomatic tibiofemoral KOA or a combined unilateral symptomatic tibiofemoral knee and hip OA.
* Clinical signs of significant effusion with noticeable swelling and/or inflammation related severe pain during the treatment visit.
* Evidence of active lymphatic or venous stasis or serious blood disorders (e.g., anemia), bleeding disorders (e.g., hemophilia), blood clots, or blood cancers (e.g., leukemia, lymphoma, and myeloma).
* Active bacterial infection, resulting in hospitalization and/or requiring intravenous antibiotic treatment.
* Synovial infection, skin infections or any skin diseases in the area of the injection site.
* History of autoimmune diseases that cause chronic joint pain and inflammation in the knee joint, including rheumatoid arthritis, psoriasis arthritis, juvenile idiopathic arthritis, systemic lupus erythematosus, gout, pseudogout, systemic sclerosis, Sjögren's disease, adult-onset still's disease.
* Known or suspected generalized chronic pain disorder.
* Severe alteration of mobility preventing any functional assessment.
* Allergy or hypersensitivity to any of the product components.
* Conditions (orthopedic, rheumatologic, musculoskeletal or inflammatory) causing symptomatic and/or radiating pain in the lower extremities that might interfere with the symptomatic OA knee pain, including hip OA assessed by physical examination by the physician.
* Symptomatic patellofemoral knee OA.
* Oral corticotherapy ≥4 mg/day (in prednisone equivalent) in the last 3 months before injection.
* Severe acute illness within 14 days prior to investigational device administration.

Any intra-articular injection (hyaluronan, hydrogel, soft implant, corticosteroid, platelet-rich plasma, local anesthetic etc.) arthroscopy, surgery in the treated knee; or cell-based therapy or an invasive procedure on the treated knee in the last 6 months before screening visit.

* Anticipated need for any surgical or other invasive procedure throughout the course of the clinical investigation, including prosthesis in the treatment knee, any concurrent OA treatments including alternative treatments (e.g., acupuncture, ultrasound, magnetic resonance etc.).
* Any investigator-assessed clinically significant condition that may represent a substantial risk to the patient or may have an impact on the study assessments.
* Participation in another clinical trial in the last 3 months before injection.
* Pregnancy and breastfeeding.
* Legal incapacity or limited legal capacity to consent.
* Trauma of the treatment knee in the last 6 months before the treatment visit.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety of Hydrogel OA 2% in subjects with symptomatic KOA | From the treatment to the end of the follow up at 26 weeks
  The primary aim of this study is to test the safety of Hydrogel OA 2% in patients with symptomatic KOA. Specifically, the aim is to demonstrate that the proportion of patients experiencing Hydrogel OA 2%-related AEs is equal to the the proportion of patients experiencing Durolane-related AEs .

SECONDARY OUTCOMES:
The improvement in the Knee Injury and Osteoarthritis Outcome Score (KOOS) 'Pain' score at 26 weeks after treatment | From the treatment to the end of the follow up at 26 weeks
  The aim is to show that the change in Knee Injury and Osteoarthritis Outcome Score (KOOS) 'Pain' score in the treatment group is at least equal to the control group at 26 weeks after treatment

OTHER OUTCOMES:
An improvement in Knee Injury and Osteoarthritis Outcome Score (KOOS) scores at 26 weeks after treatment, compared to baseline. | From the treatment to the end of the follow up at 26 weeks
  * An improvement in KOOS 'Symptoms' score compared to baseline.
  * An improvement in KOOS 'Stiffness' score compared to baseline.
  * An improvement in KOOS 'Function, Daily Living' score compared to baseline.
  * An improvement in KOOS 'Function, Sports and Recreational Activities' score compared to baseline.
  * An improvement in KOOS 'Quality of Life' score compared to baseline.
  * Change in overall KOOS score compared to baseline.

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - More Institute, Antwerp
  - AZ Sint Jan Brugge, Bruges
  - UZ Antwerpen, Edegem
  - CHU Liège, Liège
  - AZ DELTA, Roeselare

IPD SHARING:
Plan to Share IPD: No